CLINICAL TRIAL: NCT00124215
Title: A Phase 1 Double-Blind, Placebo Controlled, Dose-Escalation, Multi-center Therapeutic Trial of the Safety, Immunogenicity, and Efficacy of GI-5005; an Inactivated Recombinant Saccharomyces Cerevisiae Expressing a Hepatitis C Virus NS3-Core Fusion Protein, in Patients With Chronic Hepatitis C Infection
Brief Title: Safety and Efficacy of the Therapeutic Vaccine GI-5005 Versus Placebo for the Treatment of Chronic Hepatitis C Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlobeImmune (Industry)
Responsible Party: John Ferraro, MBA Director Clinical Operations, GlobeImmune, Inc.
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: GI-5005-01
Record Dates: First submitted 2005-07-25; First posted 2005-07-27 (Estimated); Last update posted 2010-05-05 (Estimated); Status verified 2010-05

CONDITIONS: Hepatitis C
Keywords: Hepatitis; HCV; vaccine; Hepatitis C Infection
MeSH Terms: conditions — Hepatitis C; Hepatitis | interventions — GI 5005

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

INTERVENTIONS:
Biological: GI-5005 — Heat-killed yeast cell transfected with NS3-Core fusion protien.

SUMMARY:
The GI-5005 therapeutic vaccine or placebo will be injected under the skin of hepatitis C virus (HCV) subjects. Patients will be monitored for safety, immune responses and any therapeutic benefits related to the injections.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic hepatitis C virus infection including treatment naive subjects as well as subjects who are partial responders and relapsers to prior interferon therapy
* >18 years of age
* Negative skin test for hypersensitivity to saccharomyces cerevisiae.

Exclusion Criteria:

* Non-responders to previous interferon treatments
* Cirrhosis
* HCV treatment within 3 months
* Hepatitis B infection
* HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2005-06; Primary Completion 2007-06 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 1 year

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Huntington Medical Research Institutes, Pasadena, California
  - University of Colorado Health Sciences Center, Denver, Colorado
  - University of Miami, Miami, Florida
  - University of Chicago, Chicago, Illinois
  - Weill Medical College of Cornell University, New York, New York